CLINICAL TRIAL: NCT01277276
Title: Study of Chemotherapy Side Effects in Cancer Patients: Non-invasive Optical Measurements of the Brain
Status: Withdrawn | Type: Observational
Why Stopped: no participant enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Edward L. Nelson, M.D, Associate Professor of Medicine, University of California, Irvine
Other Study IDs: 20086549
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Signs and Symptoms
Keywords: Medical tool
MeSH Terms: conditions — Signs and Symptoms | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic tool: Diffuse optical spectroscopy and Near infrared spectroscopy are non-invasive methods measure tissue hemodynamics in real time, direct quantitative information and insights treatment-associated toxicity.
  Interventions: Device: Diffuse optical spectroscopy and Near infrared spectroscopy

INTERVENTIONS:
Device: Diffuse optical spectroscopy and Near infrared spectroscopy — Diffuse optical spectroscopy and Near infrared spectroscopy are non-invasive methods measure tissue hemodynamics in real time, direct quantitative information and insights treatment-associated toxicity.

SUMMARY:
Currently there is no methodology that can assign a risk of development of chemo brain and thus, studies to understand how and why only some patients develop chemo brain along with studies of potential treatments face major hurdles. This study will define hemodynamic/optical parameters in normal individuals and cancer patients undergoing chemotherapy potentially identifying optical parameters that are associated with the development of chemo brain, leading to new insights into the origin of the chemo brain condition, and importantly potentially identifying parameters that may predict who will develop "chemo brain" in order to directing investigations of therapies.

DETAILED DESCRIPTION:
The researcher can use Non-invasive optical imaging, diffuse optical spectroscopic imaging, measure various tissues and can determine chemo brain symptoms. Near infrared diffuse optical imaging is a real-time, non-invasive technique that measures hemodynamic variations based on changes in hemoglobin oxygenation. Tissue in general and the cerebral cortex surface in particular, are transparent to near infrared light.

Direct optical measurement of cerebral hemodynamic parameters is superior to systemic approaches that infer brain levels of hemoglobin. Optical imaging in conjunction with physiologic maneuvers measures vascular tone and reactivity and may permit early detection of changes in physiology that precede the onset of chemo brain symptoms. Since chemo brain specifically impacts working memory and executive function the optical imaging can measure the frontal cortical areas behind the forehead.

ELIGIBILITY:
Inclusion Criteria:

* have a histologically proven cancer.
* Planned initiation of chemotherapy
* age range between 18-70 years

Exclusion Criteria:

* have NO a histologically proven cancer.
* NO planned chemotherapy
* age less than 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Measurement of brain tissues blood flow | 6 months
  Diffuse optical spectroscopy and Near infrared spectroscopy are non-invasive methods measure tissue hemodynamics in real time, direct quantitative information and insights treatment-associated toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nelson, MD, Principal Investigator — Beckman Laser Institute University of California Irvine; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute University of California Irvine